CLINICAL TRIAL: NCT04294602
Title: Efficacy Of Different Types Of Physiotherapy Approaches In Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Abdurrahman Tanhan, research assistant, Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BitlisErenU1
Record Dates: First submitted 2020-02-29; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Temporomandibular Disorder
Keywords: Temporomandibular disorders; Exercise; Low-level laser therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders; Motor Activity | interventions — Exercise; Low-Level Light Therapy; Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Program (Experimental): This group received therapeutic exercises and patient education. For patients to encounter fewer problems and to reduce their problems, some recommendations were made that should be taken into consideration in daily life. These suggestions were given in writing. The exercise program included muscle stretching, massage of painful muscles, guided opening and closing movements, gentle isometric tension exercises against resistance, correction of body posture and relaxation techniques. All exercises were done in 6 repetitions a set, 3 sets a day, 3 days a week, treatment program lasted 4 weeks.
  Interventions: Other: Exercise; Other: Patient Education
- Low Level Laser Therapy Program (Experimental): This group received LLLT, therapeutic exercises and patient education in the therapy programs. LLLT (max output power: 1200mW, wavelength: 808 nm, dosage: 10j/ cm2 Electronica Pagani Laser Tower Light, Italy) 2.5-4j/TrP dosage was applied to MTrP or sensitive points. The application was applied to MTrP or sensitive points in the mastication and cervical muscles.LLLT program was done in 3 days a week, the treatment program lasted 4 weeks.
  Interventions: Other: Exercise; Other: Low Level Laser Therapy; Other: Patient Education
- Manual Pressure Release Program (Experimental): ThisThis group received manual pressure release (MPR), therapeutic exercises and patient education in the therapy programs. MPR technique is a noninvasive method based on pressure on the trigger point in accordance with the patient's tolerance and technique applies supine position relax as much as possible, MTrPs in the mastication and neck muscle. Applied pressure gradually with finger over the MTrPs until the subject reported a 'moderate but easily tolerable' pain value of 7 out of 10. When the pain value decreased to at least 3 or 4 therapist increased pressure again until discomfort and/or pain appeared again. This process was repeated until there was no MTrP tension/tenderness or 60 s had elapsed. MPR program was done in 3 days a week, the treatment program lasted 4 weeks.
  Interventions: Other: Exercise; Other: Manuel Pressure Release; Other: Patient Education

INTERVENTIONS:
Other: Exercise — Exercise therapy intended in reducing muscle spasm, improving coordination of the mastication muscles and alter the jaw closure pattern.
Other: Low Level Laser Therapy — LLLT (max output power: 1200mW, wavelength: 808 nm, dosage: 10j/ cm2 Electronica Pagani Laser Tower Light, Italy) 2.5-4j/TrP dosage was applied to MTrP or sensitive points.
  Arms: Low Level Laser Therapy Program
Other: Manuel Pressure Release — MPR technique is a noninvasive method based on pressure on the trigger point in accordance with the patient's tolerance and technique applies supine position relax as much as possible, manuel pressure applied trigger point in neck and mactication muscles
  Arms: Manual Pressure Release Program
Other: Patient Education — Some suggestions were made to TMD people who should pay attention to in daily life. These suggestions were given in writing.

SUMMARY:
The aim of this study is to investigate the efficacy of different types of physiotherapy approaches in cases with cervical myofascial painful TMD.

DETAILED DESCRIPTION:
59 persons with TMD diagnosed by the dentist and with cervical myofascial pain, aged 18-30 years will be randomly allocated, 3 groups. The participants were randomly allocated only exercise group (EG) (n=20), low-level laser therapy plus exercise group (LLLT) (n=17) and manual pressure release plus exercise group (MPR) (n=22). The cases were evaluated and treated by the same physiotherapist for 4 weeks (12 sessions).

Pain, pain pressure threshold, temporomandibular joint (TMJ) mobility and disability, forward head posture, head rotation, neck disability, psychological status and quality of life were evaluated. Evaluations were repeated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cases who have 3 or more symptoms related to TMJ problems
* cases who have trigger points in cervical and masticatory muscles
* cases who TMD detected by the dentist,
* being between the ages of 18-30,
* volunteer to participate in the study

Exclusion Criteria:

* Patients with a positive history of trauma in the face and neck area and neurological disorders
* patients undergoing TMJ or cervical region surgery in the last 3 months,
* patients who used dental orthotics within 1 month,
* patients who have TMJ instability,
* patients who have cervical and upper thoracic region,
* patients who have active infection and chronic pain, such as trigeminal neuralgia

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold Assessment | Change from baseline pressure pain threshold score in neck and mastication muscles at week 4.
  Pressure Pain Threshold (PPT) of an individual's mastication and cervical muscle was measured with an algometer (JTECH Medical Industries, CommanderTMAlgometer), and the applied pressure was increased to 1 cm2/ kg per second. PPT measurements were repeated three times and the average was used for analysis in every participant.
Pain Severity Assessment | Change from baseline TMJ pain and intensity of head pain, TMJ noise and jaw locking score at week 4.
  To evaluate the general pain severity of the patients, the Visual Analog Scale (VAS), which is the Visual Pain Scale of Turkish, was used. Patients were asked to mark their general pain separately on a 10 cm scale. According to this, "0" indicates that there is no pain, and "10" indicates the most severe pain. The distance between the marked point and the beginning of the line was recorded in centimeters
Jaw Movements Assessment | Change from baseline MMO and lateral deviation score at week 4.
  Maximum mouth opening (MMO) and lateral deviation were measured with a caliper.
Neck Movements Assessment | Change from baseline cervical rotations and craniovertebral angle score at week 4.
  Cervical rotations and the craniovertebral angle between C7 and tragus were measured by a goniometer.
Temporomandibular Disorder Severity | Change from baseline temporomandibular disorder severity score at week 4
  The TMD severity in participation is defined by the Craniomandibular Index (CMI) which was developed to provide a standardized measure to the severity of problems in mandibular movement, muscle, and joint tenderness and TMJ noise for use in epidemiological and clinical outcome studies. The instrument was designed to have clearly defined objective criteria, simple clinical methods, and ease in scoring; it is divided into the Palpation Index (PI) and the Dysfunction Index (DI). The means of the subscales were averaged to produce a CMI score ranging from 0 (best) to 1 (worst)
Quality of Life Assesment | Change from baseline quality of life score at week 4
  Short Form-36 questionnaire contains the physical and mental component, which is evaluated, is close to 100, indicating an increase in health-related quality of life. The means SF-36 score ranging from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Neck Disability Assesment | Change from baseline neck disability score at week 4.
  Northwick Park Neck Pain Questionnaire; Neck pain severity, neck pain and sleep, numbness and tingling in the arms at night, duration of symptoms and complaints, weight-bearing, reading and watching television, work and housework, social activities and driving includes 9 items. Each item consists of 5 options, the level of disability increases as you approach 36 points. The means northwick park neck pain questionnaire score ranging from 0 (best) to 36 (worst).
Psychological Status Assesment | Change from baseline psychological status score at week 4.
  Beck depression index which is a two-factor scale, emotion and somatic, has 21 questions, the lowest score is 0 and the highest score is 3 in each question. The means Beck depression index score ranging from 0 (best) to 63 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Abdurrahman TANHAN, MSc, Principal Investigator — Bitlis Eren University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)